CLINICAL TRIAL: NCT06629961
Title: Impact of Connection and Disconnection of the Transepithelial Abutment in Dental Implants
Brief Title: Impact of Transepithelial Abutment Connection and Disconnection in Dental Implants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, David Peñarrocha Oltra, Associate Professor of Stomatology, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3395885
Record Dates: First submitted 2024-07-31; First posted 2024-10-08 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Bone Loss; Bacterium; Agent; Satisfaction, Patient
Keywords: bone loss; bacteria; dental implant; satisfaction
MeSH Terms: conditions — Bone Diseases, Metabolic; Patient Satisfaction; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abutment Group (Experimental): The patients in this group will undergo implant placement surgery using the conventional technique, which will include a full-thickness flap, biological drilling, and sub-crestal implant placement at 2 mm below the crest level. Since this is the Pilar group (Galimplant aesthetic straight abutment, NUEVAGALIMPANT), a 3 mm abutment will be placed during the same procedure, secured with a torque of 30 N. A healing cap will be applied and maintained until the osseointegration process is completed after three months.
  After three months, this group will receive a cement-retained and screw-retained zirconia prosthesis, which will be placed over the previously installed abutment. The crown screw will be torqued to 25 N.
  Interventions: Procedure: abutment placement
- ti-base Group (Experimental): The patients in this group will undergo implant placement surgery using the conventional technique, which will include a full-thickness flap, biological drilling, and sub-crestal implant placement at 2 mm below the crest level. Since this is the Tibase group (3 mm Tibase from Galimplant, NUEVAGALIMPANT), submerged healing will be performed with a healing cap connected to the implant, which will remain in place until the osseointegration process is completed after three months.
  After three months of osseointegration, a prosthesis will be placed directly connected to the implant platform via the 3 mm Tibase. The screw will be tightened to 30 N.
  Interventions: Procedure: Ti-base placement

INTERVENTIONS:
Procedure: abutment placement — Placement of a subcrestal implant at more than 35 N and placement of a trans-epithelial abutment at 30 N
  Arms: Abutment Group
Procedure: Ti-base placement — Placement of a subcrestal implant at more than 35 N and placement of a Tibase placement at 30 N
  Arms: ti-base Group

SUMMARY:
Over the past decade, implant research has focused on maintaining the health and stability of peri-implant tissues. A key factor is platform switching at the bone level, where a narrower abutment than the implant is used. This technique increases the implant's horizontal surface area for biological width establishment and reduces stress on the crestal bone.

Studies showed that repeated disconnection and reconnection of prosthetic components could compromise the mucosal barrier around implants, leading to an apical shift in the connective tissue junction and vertical tissue loss. This led to the "one abutment, one time" protocol, advocating the placement of the definitive abutment during initial implant surgery to avoid its removal during healing.

A recent meta-analysis indicated bone loss at the marginal level due to abutment connection and disconnection, despite different treatment protocols. Thus, a standardized abutment between the fixed prosthesis and the implant has been recommended to preserve marginal bone levels. This approach moves the biological width apically, protecting the bone from irritation and improving marginal bone isolation.

However, comparative evidence between direct implant-connected prostheses and trans-epithelial abutments is lacking. This study aims to evaluate the "one abutment, one time" protocol's effect on bone loss 12 months after prosthesis placement.

Secondary objectives include assessing patient satisfaction using Patient-Reported Outcome Measures (PROM) during prosthesis fabrication and placement, and obtaining information on the diversity and function of microorganisms on the implant using metagenomic techniques 12 months post-prosthesis placement.

Throughout the prosthesis fabrication and the first 12 months, various evaluations will be conducted in both abutment and Ti-base groups:

* **Bleeding:** Recorded during various prosthetic stages.
* **Pain:** Assessed using a visual analog scale after each stage.
* **Anesthesia:** Recorded if used at each stage.
* **Radiographs:** Number taken to check the fit.
* **Time:** Measured for each prosthetic phase.
* **Repetitions:** Number of repeated procedures quantified.
* **Metagenomic tests:** Samples collected following the Human Microbiome Project protocol to analyze microbial diversity and function.

ELIGIBILITY:
Inclusion Criteria:

* Healthy partially edentulous adult patients needing at least two implants for the placement of single or consecutive crowns in the posterior mandible or maxilla will be recruited.
* These patients should exhibit a plaque index and gingival bleeding index of less than 25%, and have sufficient bone height and width for the placement of dental implants measuring 8 or 10 mm in length and 3.5 or 4 mm in diameter.
* Additionally, they must have at least 2 mm of keratinized vestibular gingiva, stable occlusion, and a periodontium in good health

Exclusion Criteria:

* Edentulous areas requiring bone grafts will be excluded.
* Patients with medical conditions contraindicating implant surgery, such as severe bruxism or inadequate oral hygiene.
* Pregnant or lactating women, patients undergoing bisphosphonate therapy, those receiving chemotherapy or radiotherapy in the head and neck area, non-compliant patients with incomplete data records, and those who do not attend regular follow-up appointments will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
periimplant marginal bone loss | 12 months
  The peri-implant marginal bone level was measured using Image J software from the National Institutes of Health with an accuracy of 0.1 mm. A straight line was drawn at the implant platform level (representing zero height), and perpendicular lines were drawn from the mesial and distal sides of the platform to measure the distance to the bone level on each side

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Clínica Odontológica de la Universitat de Valencia, Fundación Lluis Alcanyis, Valencia
  - Facultad de Medicina y Odontología de la Universitat de València, Valencia